CLINICAL TRIAL: NCT02248935
Title: Prospective Cohort Study Comparing Two Lightweight Y Meshes After Robotic-Assisted Laparoscopic Sacrocolpopexy Longterm Outcomes
Brief Title: Comparison of 2 Lightweight Y-meshes After Laparoscopic Sacrocolpopexy
Status: Completed | Type: Observational
Sponsor: Atlantic Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 599819-2
Record Dates: First submitted 2014-08-25; First posted 2014-09-25 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Pelvic Organ Prolapse
Keywords: Robotic Assisted Laparoscopic Sacrocolpopexy; Y Mesh; Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Repair with Alyte or Restorelle Y-Mesh: Women who underwent their index robotic-assisted laparoscopic sacrocolpopexy at Morristown Medical Center or Overlook Medical Center using either the Alyte Y-mesh or Restorelle Y-smartmesh between 1/2007 and 8/2011.

SUMMARY:
The purpose of the study is to determine the clinical cure rates of pelvic organ prolapse from subjects that had a robotic-assisted sacrocolpopexy using Alyte Y mesh and Restorelle Y smartmesh lightweight mesh.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent robotic-assisted laparoscopic sacrocolpopexy between January 2007 to August 2011 using either Alyte Y-mesh or Restorelle Y-mesh

Exclusion Criteria:

* Refusal to participate in our long-term outcome study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women who had a robotic-assisted laparoscopic sacrocolpopexy using either mentioned Y-mesh during the listed timeframe. All of the index cases were performed by fellowship-trained FPMRS specialists.
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Clinical Cure Rate | 5-6 years
  To be considered a "clinical cure" subjects must meet all of the following criteria: no re-operation for or non-surgical treatment of pelvic organ prolapse since the index surgery; no symptoms of vaginal bulge as measured by a validated symptom questionnaire; no Pelvic Organ Prolapse Quantification (POP-Q) points greater than 0; POP-Q point C less than or equal to -5; an answer of "satisfied" or "very satisfied" on validated Surgical Satisfaction Questionnaire

SECONDARY OUTCOMES:
Objective Anatomic Outcome | 5-6 year
  POP-Q measurements of Pelvic Organ Prolapse will be measured comparing both mesh groups and entire combined cohort compared to 12 month findings
Mesh exposure/erosion | 5-6 years
  The rate of mesh exposure or erosion will be measured
Complications | 5-6 years
  any other complications related to the index surgery will be documented
Symptom Comparison | 5-6 years
  to compare related symptoms such as urinary frequency, bowel function, and sexual function both between mesh groups and for the entire group compared to 12 month findings
Surgical Satisfaction | 5-6 years
  The validated Surgical Satisfaction Questionnaire will be used to measure overall surgical satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urogynecology-Atlantic Health System, Morristown, New Jersey, United States

REFERENCES:
- [Derived] Culligan PJ, Lewis C, Priestley J, Mushonga N. Long-Term Outcomes of Robotic-Assisted Laparoscopic Sacrocolpopexy Using Lightweight Y-Mesh. Female Pelvic Med Reconstr Surg. 2020 Mar;26(3):202-206. doi: 10.1097/SPV.0000000000000788. PMID 31688526